CLINICAL TRIAL: NCT01900730
Title: Randomized Phase II Double Blind Study of Valproic Acid (VPA) vs Placebo to Shorten Time of Indwelling Pleural Catheter
Brief Title: Study of Valproic Acid (VPA) vs Placebo to Shorten Time of Indwelling Pleural Catheter
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Inflammatory Breast Cancer Network Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0930; NCI-2014-01196 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Metastatic; Indwelling pleural catheter; Valproic acid; VPA; Depakene; Placebo; Pill diary; Drainage diary; Questionnaires; Surveys
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Valproic Acid; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patient takes placebo capsule 3 times a day by mouth for 10 weeks. Patient contacted by phone to assess tolerance and instruction to increase dose. Questionnaires completed at baseline, weeks 2, 6, and 10. Patient given a pill diary to record the time each dose taken. Patient completes daily diary of drainage with the date and amount of fluid drained each day at home. Drained fluid from the day before brought to each clinic visit to give to the research team.
  Interventions: Drug: Placebo; Behavioral: Questionnaires; Behavioral: Pill Diary; Behavioral: Drainage Diary
- Valproic Acid (VPA) (Experimental): Patients initially receive daily oral VPA 15 mg/kg/day divided in three doses. If patient tolerates the reduced dose for 10 consecutive days, then the VPA dose will increase to 30 mg/kg/day divided into three doses. Patients treated for 10 weeks. Questionnaires completed at baseline, weeks 2, 6, and 10. Patient given a pill diary to record the time each dose taken. Patient completes daily diary of drainage with the date and amount of fluid drained each day at home. Drained fluid from the day before brought to each clinic visit to give to the research team.
  Interventions: Drug: Valproic Acid (VPA); Behavioral: Questionnaires; Behavioral: Pill Diary; Behavioral: Drainage Diary

INTERVENTIONS:
Drug: Placebo — Patient takes placebo capsule 3 times a day by mouth for 10 weeks.
  Arms: Placebo
Drug: Valproic Acid (VPA) — Patients initially receive daily oral VPA 15 mg/kg/day divided in three doses. If patient tolerates the reduced dose for 10 consecutive days, then the VPA dose will increase to 30 mg/kg/day divided into three doses. Patients treated for 10 weeks.
  Other Names: Depakene
  Arms: Valproic Acid (VPA)
Behavioral: Questionnaires — Questionnaires completed at baseline, weeks 2, 6, and 10.
  Other Names: Surveys
Behavioral: Pill Diary — Patient given a pill diary to record the time each dose taken.
Behavioral: Drainage Diary — Patient completes daily diary of drainage with the date and amount of fluid drained each day at home. Drained fluid from the day before brought to each clinic visit to give to the research team.

SUMMARY:
The goal of this clinical research study is to learn if receiving valproic acid (VPA) compared to a placebo can reduce the amount of time you will need to have an indwelling pleural catheter compared to the standard of care, which involves using an indwelling pleural catheter alone.

VPA is designed to stop cancer cells from dividing and maturing. This may cause the cancer cells to become less malignant and cause less pleural fluid production.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Baseline Fluid Collection:

Before receiving the study drug or the placebo, pleural fluid will be drained from your catheter to be compared to fluid collected later in the study.

Study Groups:

You will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups.

Group 1 will take a placebo 3 times a day for 10 weeks while an indwelling pleural catheter drains pleural fluid.

If you are in Group 2, you will take VPA 3 times a day for a total of 10 weeks while an indwelling pleural catheter drains pleural fluid.

Study Drug Administration:

Within 48 hours of collection of baseline fluid, all study participants will take either placebo or VPA capsules 3 times a day by mouth with food. If you tolerate the starting dose well and the study doctor thinks it is in your best interest, your dose level will be doubled. You may be contacted at a later time by telephone to discuss how you are doing with the medicine. If your doctor feels your dose should be doubled, he/she will talk to you about it at this time.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

You will be given a pill diary to record the time you take each dose. You will need to bring the diary with you to every clinic visit.

The fluid drained from the catheter will be collected and studied to see if the how the VPA is working and how it may affect the time you will need to have an indwelling pleural catheter.

You will also be asked to keep a daily diary of drainage with the date and amount of fluid drained each day at home. You will bring the drained fluid from the day before to each clinic visit to give to the research team. You will be given special containers to store the drained fluid. You will only save fluid from the day before each clinic visit. On the other days you will write down the amount of drained fluid that was collected, then you can throw away the fluid. You must bring the daily drainage diary to each clinic visit.

Study Visits:

At Weeks 2, 6, and 10 while you are receiving the study drug:

* You will have a complete physical exam including weight and vital signs and a medical history.
* You will complete the same questionnaires that you completed at screening.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a chest X-ray to check the status of the disease.

At Week 10 only, you will have a computed tomography (CT) scan of the chest to check the status of the disease.

Length of Study:

You will be taken off study after the indwelling pleural catheter has been removed. You will no longer be able to take part in this study if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions. Your active participation in this study will be over after Week 10.

Follow-Up Medical Record Review:

After the 10 week visit the study personnel will continue to review your medical record to learn when the indwelling pleural catheter was removed. Your medical record information will continue to be reviewed for up to 5 years.

This is an investigational study. VPA is FDA approved and commercially available for the treatment of epileptic seizures and mania in bipolar disorder. VPA use in patients using pleural catheters is for research purposes only.

Up to 76 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic pleural effusion requiring the presence of an IPC or new placement of an IPC.
2. Pathologic documentation of breast cancer.
3. Performance status 0 to 3 (ECOG scale).
4. Signed informed consent.
5. Subject must be female or male age 18 years or over.
6. At least one prior line of chemotherapy in the metastatic setting.
7. Positive effusion cytology.

Exclusion Criteria:

1. Other prior malignancy (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer) from which the patient has been disease-free for at least two years.
2. Laboratory results sustained at: Neutrophils less than 1.5 × 109/L ; Serum bilirubin >1.5 x the upper limit of reference range (ULRR); Serum creatinine >1.5 x ULRR or creatinine clearance < 30 mL/minute (calculated by Cockcroft-Gault formula).
3. Patients with a history of existing hypercalcemia, hypocalcemia, hypermagnesemia or hypomagnesemia that is not corrected despite supplementation. Known Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × ULRR or alkaline phosphatase (ALP) >2 x ULRR, or > 4x ULRR if judged by the investigator to be related to liver metastases.
4. Serious underlying medical condition that would impair the ability of the patient to receive protocol treatment, specifically cardiac diseases, uncontrolled hypertension or renal diseases.
5. Diagnosis of an infection requiring IV antibiotics 14 days prior to registration.
6. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
7. Women who are currently pregnant or breast feeding.
8. Known hypersensitivity to VPA, valproate sodium, disodium valproate, or any ingredient in the respective formulation.
9. Known urea cycle disorders based on history.
10. Known HIV infection based on history.
11. Active or recent pancreatitis (within last 6 months).
12. Any of the following interventions on the affected hemithorax: prior IPC, prior chest tube placement, history of chemical or mechanical pleurodesis, history of thoracotomy within 4 weeks and incompletely healed surgical incision before randomization.
13. Evidence of empyema or history of empyema of the affected hemithorax.
14. Non-correctable bleeding diathesis.
15. Clinical evidence of skin infection at the potential site of IPC placement.
16. Patients currently taking valproic acid.
17. History of hepatitis or liver disease.
18. The following drugs will not be administered concurrently with VPA: Carbapenem antibiotics; Clonazepam; Topiramate; Felbamate; Lorazepam; Barbiturates; Barbiturates; CarBAMazepine; ChlorproMAZINE; Ethosuximide; GuanFACINE; LamoTRIgine; MethylfolateOXcarbazepine; Paliperidone; Phenytoin; Primidone; Protease Inhibitors; Rifampin; Risperidone; Rufinamide; Salicylates; Temozolomide; Tricyclic Antidepressants; Vorinostat; Zidovudine.
19. History of seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy A. Woodward, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 3 participants started, only 1 completed with the other 2 withdrawing before treatment. The protocol was terminated early due.
Pre-assignment Details: All participants are listed in Group 1 due to this is a double blinded study and unable to determine which groups the participants were enrolled on.
Groups:
- Group 1: Group 1 will take placebo 3 times a day for 10 weeks while an indwelling pleural catheter drains pleural fluid.
- Group 2: Group 2 will take valproic acid (VPA) 3 times a day for a total of 10 weeks while an indwelling pleural catheter drains pleural fluid.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 3 | 0
Completed | 1 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Screen Failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early with low accrual.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Pleural Catheter Removal
Description: Primary outcome is time to pleural catheter removal because it is no longer needed to drain the pleura of fluid. Time to catheter removal measured from the date of placement of the catheter to the date it is removed. Cox (1972) proportional hazards regression used to model time to catheter removal as a function of treatment arm, cytology, and lung re-expansion, as well as other potential prognostic factors, including ECOG performance status, number of circulating tumor cells in peripheral blood and in pleural effusion.
Time Frame: 10 weeks
Population: Study terminated early with single patient leaving low accrual with insufficient data for analysis
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of registration through study completion and follow up, assessed up to 5 years
Description: Of the 3 participants started, only 1 completed with the other 2 withdrawing before treatment 1 withdrew and 1 screen failure. The protocol was terminated early.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=1) | Group 2 (N=0)
Urinary frequency (Renal and urinary disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT01900730/Prot_SAP_000.pdf